CLINICAL TRIAL: NCT02870686
Title: A Prospective Randomized Trial Comparing EUS Guided ERCP Without Fluoroscopy With Standard ERCP in Common Bile Duct Stone Removal
Brief Title: EUS Guided ERCP in Bile Duct Stone Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Nisa Netinatsunton, Principal Investigator, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC: 56-199-21-3-2
Record Dates: First submitted 2016-08-13; First posted 2016-08-17 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-06

CONDITIONS: Choledocholithiasis
Keywords: ERCP; EUS guided ERCP without fluoroscopy
MeSH Terms: conditions — Choledocholithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ERCP without the use of fluoroscopy (Active Comparator): Patients with uncomplicated bile duct stones detected by EUS was assigned to the EUS guided ERCP without fluoroscopy clear all of the bile duct stones.
  Interventions: Procedure: ERCP without the use of fluoroscopy
- ERCP with the use of fluoroscopy (Active Comparator): Patients with uncomplicated bile duct stones detected by EUS was assigned to underwent ERCP with the use of fluoroscopy to clear all of the bile duct stones.
  Interventions: Procedure: ERCP with the use of fluoroscopy

INTERVENTIONS:
Procedure: ERCP without the use of fluoroscopy — ERCP removal of stone technique without the use of fluoroscopy involves: (1) catheter with wire achieve bile duct, (2) confirmation of bile duct achievement with catheter aspiration of bile, (3) performance of endoscopic biliary sphinctertome, (4) stone removal with balloon or basket- number of stones removed should compare number detected on EUS, (5) confirmation of complete stone clearance with radiocontrast.
  Arms: ERCP without the use of fluoroscopy
Procedure: ERCP with the use of fluoroscopy — ERCP removal of stone technique with the use of fluoroscopy involves: (1) catheter with wire achieve bile duct, (2) confirmation of bile duct achievement with fluoroscopy images, (3) performance of endoscopic biliary sphinctertome, (4) stone removal with balloon or basket, (5) confirmation of complete stone clearance with radiocontrast.
  Arms: ERCP with the use of fluoroscopy

SUMMARY:
For endoscopist, ERCP for bile duct stone removal is the most widely performed procedure. However, the risk associated radiation exposure to patients and staff are not neglible. Earlier studies, ERCP without the use of fluoroscopy has been reported high success for bile duct stone removal in pregnant patients to prevent radiation exposure to the fetus. EUS is highy accurate technique in detecting common bile duct stone and guiding for therapeutic intervention. There has been a few data from literature showed that EUS guided CBD stone ( CBDS ) removal are equivalent to those following ERCP in term of successful CBDS removal and complications. This randomized trial is designed to address the question that EUS guided CBDS removal is equivalent to ERCP in term of efficacy and safety.

DETAILED DESCRIPTION:
Common bile duct stones (CBDS) can be complicated with various conditions including biliary pain, acute cholangitis, acute pancreatitis and secondary biliary cirrhosis. CBDS should therefore be removed even if patients are asymptomatic.

Endoscopic retrograde cholangiopancreatography (ERCP) is the cornerstone treatment of CBDS. ERCP is often performed under fluoroscopic guidance. This comprises biliary cannulation whereby the bile duct is achieved with a standard ERCP catheter under fluoroscopy guidance, radiocontrast was injected for confirmation and images of biliary system, location and number of CBDS, biliary sphincterotomy was then performed followed by stone extraction using a standard accessories such as a basket and or balloon. Therefore, the endoscopist, endoscopic staff and patient are potentially exposed to ionizing radiation during ERCP. Endoscopists should always attempt to minimize radiation exposure to the personnel staffs and patients by following the ALARA principle ("As Low As Reasonably Achievable"). ERCP without the use of fluoroscopy is the one method to avoid exposure to radiation. A few retrospective case series have been shown that ERCP can be performed with high success rate without the need for fluoroscopic imaging.

EUS has been proven to have diagnostic accuracy comparable to ERCP in the diagnosis of CBDS, and it's associated with a very low procedure related complications and non-radiation exposure procedure. With EUS performed before ERCP, unnecessary ERCP and its related complications can be avoided in patients without CBDS. In patients with CBDS, the images of pancreaticobiliary tract derived from EUS provide an information regarding the location, size and number of CBDS for guiding therapeutic endoscopy, and allowing a therapeutic ERCP in the same session of sedation. Vohra et al. reported the retrospective case series of EUS - based ERCP in 10 pregnant patients, they have shown that EUS performed prior ERCP can eliminate unnecessary ERCP and achieve in CBDS clearance without the use of fluoroscopy. We have previously reported the use of EUS guided ERCP in the removal of CBDS without fluoroscopy (EGWF) in the pilot study, it showed that EGWF was feasible in selected patients with CBDS. The efficacy of EUS guided ERCP in CBDS removal without fluoroscopy compared with standard ERCP has not been fully assessed. We therefore prospectively investigated the efficacy and safety of EGWF versus ERCP in CBDS removal in a larger patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had EUS presence of CBDS ≤ 10 mm, and EUS images absence of CBD stricture and CBD narrowing below the stones

Exclusion Criteria:

* pregnancy
* concomitant intrahepatic bile duct stones
* malignant bile duct stricture
* altered gastrointestinal anatomy
* instability hemodynamics
* concomitant emergency situation
* unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-05; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Treatment success | 24 months
  The number of patients who achieved complete stone clearance in either EGWF or ERCP techniques.

SECONDARY OUTCOMES:
Technical success | 24 hours
  The number of patient in whom bile duct was accessed with guide wire in either EGWF or ERCP techniques.

OTHER OUTCOMES:
Compare procedure time | 24 hours
  Compare procedure time defined as the time between insertion of the catheter and the final occlusion cholangiogram in either EGWF or ERCP groups.
Compare fluoroscopy time | 24 hours
  Compare fluoroscopy time defined as the total time of using of fluoroscopy in performing procedure in either EGWF or ERCP groups.
Complication rate | 30 days
  The number of patients who developed complications related procedure included pancreatitis, bleeding, perforation, cholangitis as defined and graded according to the consensus guideline and sedation related complications in either EGWF or ERCP techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Nisa Netinatsunton, MD., Principal Investigator — NKC Institute of Gastroenterology and Hepatology , Faculty of Medicine, Prince of Songkla University.
Locations (1):
- NKC Institues of Gastroenterology and Hepatology, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No
The individual data of patients participating in the study are not available for public sharing since we did not obtain the consent to share the data of patient

REFERENCES:
- [Derived] Netinatsunton N, Sottisuporn J, Attasaranya S, Witeerungrot T, Siripun A, Pattarapuntakul T, Ovartlarnporn B. Prospective randomized trial of EUS-assisted ERCP without fluoroscopy versus ERCP in common bile duct stones. Gastrointest Endosc. 2017 Dec;86(6):1059-1065. doi: 10.1016/j.gie.2017.03.1539. Epub 2017 Apr 7. PMID 28392365